CLINICAL TRIAL: NCT00379925
Title: A Partnership to Promote Physical Activity and Healthy Eating in AME Churches
Brief Title: Effectiveness of a Church-Based Program at Increasing Physical Activity and Healthy Dietary Habits in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sara Wilcox, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00005414; R01HL083858 (NIH); R01HL083858-01 (NIH)
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: Physical Activity; Exercise; Dietary Habits
MeSH Terms: conditions — Obesity; Motor Activity; Feeding Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral (Experimental): Participants will take part in the Physical Activity and Dietary Health Promotion Program.
  Interventions: Behavioral: Physical Activity and Dietary Health Promotion Program
- Delayed intervention (No Intervention): Participants are assigned to a delayed intervention group and serve as a no-intervention control group.

INTERVENTIONS:
Behavioral: Physical Activity and Dietary Health Promotion Program — Churches within the intervention group will receive a committee training and church cook training designed to teach them how to do a self-assessment of current practices and develop a plan for their program. The intervention is based on the structural model of health behavior and targets opportunities, mass media (within the church), guidelines and policies, and church environment. Intervention churches also receive monthly intervention mailings to support intervention implementation.
  Arms: Behavioral

SUMMARY:
Obese African Americans are at risk for diseases such as diabetes, cancer, and heart disease. Church-based interventions have the potential to positively influence the health habits and behaviors of a large percentage of African Americans. The purpose of this study is to evaluate the effectiveness of a church-based program that emphasizes increased physical activity and healthy dietary habits among members of predominately African American churches in South Carolina.

DETAILED DESCRIPTION:
Many obesity-related diseases, including diabetes, cancer, and heart disease, occur more frequently in ethnic minorities than in Caucasians. African Americans have an extremely high church attendance rate, making church-based interventions a viable method to reach a wide audience and positively influence health habits and behaviors. The most effective way to prevent or reverse the effects of obesity is through weight loss, which can be accomplished by increasing physical activity and following a low fat and low sodium diet that emphasizes fruits, vegetables, and whole grains. Few programs have been developed that have specifically examined the effects of a church-based physical activity and dietary intervention. This study will encourage church leaders to assist in the development of a health promotion program that will incorporate the church's social, cultural, and policy influences. The purpose of the study is to evaluate the effectiveness of the intervention on increasing physical activity, improving blood pressure levels, and promoting healthy dietary habits among church members. The importance of pastor support and participation will be evaluated, and the results from this study may be used to develop additional church-based interventions across a larger geographic area.

In Year 1 of this 5-year study, representatives from the Palmetto Conference of the African Methodist Episcopal (AME) Church and three state universities in South Carolina will participate in monthly planning sessions to develop the intervention. Local health committees and church pastors and cooks will be trained to implement the program. The 18-month intervention will occur in three waves; where at least 60 churches will be randomly assigned to participate in either the immediate intervention or delayed intervention. The program will emphasize increased physical activity and the adaptation of a healthy diet that includes low fat and low sodium foods, fruits, vegetables, and whole grains. At baseline and Month 18, blood pressure will be measured, and physical activity levels and fruit and vegetable intake will be assessed for some church members. Additionally, throughout the study, some participants will wear an accelerometer, which is a small device that measures physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Member of a church in the Palmetto Conference of the 7th Episcopal District of the AME Church
* Attends church services or events at least once per month

Exclusion Criteria:

* Planning to move in the 18 months following study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2006-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 15 months
  Systolic and diastolic blood pressure
Physical activity (measured with the Community Healthy Activities Model Program For Seniors [CHAMPS] questionnaire) | 15 months
  Self-report measure of physical activity
Fruit and vegetable consumption (measured with NCI screener & 2-item measure) | 15 months
  self-report measure of physical activity

SECONDARY OUTCOMES:
Physical activity (measured with an accelerometer) | 15 months
  Accelerometer measured physical activity
Fat consumption | 15 months
  Self-reported measure of practices associated with fat consumption
Fiber consumption | 15 months
  Self-reported measure of practices associated with fiberconsumption

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wilcox, PhD, Principal Investigator — University of South Carolina
Locations (1):
- African Methodist Episcopal Churches in South Carolina, Lane, South Carolina, United States

REFERENCES:
- [Derived] Kyryliuk R, Baruth M, Wilcox S. Predictors of Weight Loss for African-American Women in the Faith, Activity, and Nutrition (FAN) Study. J Phys Act Health. 2015 May;12(5):659-65. doi: 10.1123/jpah.2013-0220. Epub 2014 Jun 4. PMID 24905567
- [Derived] Saunders RP, Wilcox S, Baruth M, Dowda M. Process evaluation methods, implementation fidelity results and relationship to physical activity and healthy eating in the Faith, Activity, and Nutrition (FAN) study. Eval Program Plann. 2014 Apr;43:93-102. doi: 10.1016/j.evalprogplan.2013.11.003. Epub 2013 Dec 10. PMID 24394548
- [Derived] Wilcox S, Parrott A, Baruth M, Laken M, Condrasky M, Saunders R, Dowda M, Evans R, Addy C, Warren TY, Kinnard D, Zimmerman L. The Faith, Activity, and Nutrition program: a randomized controlled trial in African-American churches. Am J Prev Med. 2013 Feb;44(2):122-31. doi: 10.1016/j.amepre.2012.09.062. PMID 23332327